CLINICAL TRIAL: NCT02545894
Title: An Investigation Into the Effect of a Novel, Non Verbal, Cognitive Treatment on Functional Communication in Global Aphasia
Brief Title: An Evaluation of a New Nonverbal Treatment for Global Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 13/0581
Record Dates: First submitted 2015-06-22; First posted 2015-09-10 (Estimated); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Cognitive Behavioral Therapy

ARMS (3):
- BASELINE TESTING (No Intervention): Language and cognitive assessments conducted
- Treatment (Experimental): Intervention given:
  visual tracking pressing a button every time a picture is seen on the screen
  * playing dominoes and snap
  * pressing a button every time a specific picture is seen on the screen
  * Pressing a button every time a specific sound is heard
  * Matching objects to a picture
  * Matching gestures to objects
  * Matching two connected objects
  * Sorting objects by categories
  * Matching sounds to objects
  * "Complete the category" and "odd on out with objects"
  * Choosing target objects by pointing
  * Choosing objects to complete the category by pointing
  Interventions: Behavioral: Cognitive therapy
- Post intervention (No Intervention): Repeated testing

INTERVENTIONS:
Behavioral: Cognitive therapy — The tasks are:
  * visually tracking a picture as it moves across the computer screen
  * pressing a button every time a picture is seen on the screen
  * pressing a button every time a specific picture is seen on the screen
  * Pressing a button every time a specific sound is heard
  * Matching objects to a picture
  * Matching gestures to objects
  * Matching two connected objects
  * Sorting objects by categories
  * Matching sounds to objects
  * "Complete the category" and "odd on out with objects"
  * Choosing target objects by pointing
  * Choosing objects to complete the category by pointing
  Arms: Treatment

SUMMARY:
People with global aphasia (PwGA) post stroke have little to no meaningful communication abilities (ie limited comprehension, spoken language, reading and writing abilities).A proportion of PwGA will also have limited abilities to use any alternative means of communication e.g. gesture, pictures or computer devices. There is a suggestion in the literature that this is because of co-occurring cognitive deficits. The consequence is that these clients are unable to reliably communicate even their basic needs.This is commonly known as having no functional communication abilities. Such PwGA tend not to respond to standard speech and language therapy interventions.

This research will investigate the effect of a new cognitive intervention designed to improve basic functional communication abilities. The treatment will be nonverbal and involve computer and paperbased tasks ordered hierarchically from basic to more complex tasks. Six to eight participants will take part. All their sessions will take place in their own home. For some this may be a care home. They will first complete a diagnostic communication assessment in order for baseline abilities to be established. Further formal language and cognitive assessments will be conducted over a period of 6 weeks. A relative/friend will complete a questionnaires about mood/communication. The PwGA will also be videoed interacting with the research student e.g. looking at a magazine, completing a jigsaw, answering questions and making choices non-verbally.

The participants then receive the new intervention 3 times a week for 6 consecutive weeks. All intervention sessions will be videoed. Then participants will be reassessed over 2 weeks using the same assessments as prior to the intervention. The questionnaire with their relative/friend and videoed activity session will also be repeated. After a twelve week break the participant will be videoed interacting with the research student complete some of the assessments again and their relative will re-complete the questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* have global aphasia as diagnosed by an SLT
* have little or no verbal output
* inconsistent single word comprehension
* little or no ability to read or write
* little or no ability to use alternative modes of communication
* Little or no ability to make choices in function
* no diagnosis/history of a progressive neurological condition
* no diagnosis of hearing loss
* no diagnosis/history of a mental health condition
* English as a first language

Exclusion Criteria:

* has another form of aphasia
* is able to consistently express basic needs non-verbally or verbally.
* is able to participate in communicative interaction with a familiar other
* has a history of a progressive neurological condition
* has hearing loss
* has a diagnosis/history of a mental health condition
* does not have English as a first language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
American Speech and Hearing Association -Functional Assessment of Communication | 27 weeks
  Questionnaire completed by friend/relative
Constructed Interaction Task | 27 weeks
  video recorded interaction

SECONDARY OUTCOMES:
Aphasia Screening Test | 14 weeks
  Language assessment
Mood Screen | 27 weeks
  depression screening tool
Pyramids and Palm Trees Test | 27 weeks
  pictorial semantic assessment
Wisconsin Card Sorting Test | 14 weeks
  cognitive assessment
Butt Non verbal reasoning test | 27 weeks
  cognitive assessment
Western Aphasia Battery cognitive sub test | 14 weeks
  cognitive assessment

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Beeke, PhD, Principal Investigator — UCL
Locations (1):
- University College London, Research Dept of Language and Cognition, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No